CLINICAL TRIAL: NCT06456359
Title: Pasireotide as Maintenance Treatment With Monthly Deep Intramuscular Injection in SSTR2/3/5-Expressing Synovial Sarcoma and Desmoplastic Small Round Cell Tumor
Brief Title: Pasireotide as Maintenance Treatment in Synovial Sarcoma and Desmoplastic Small Round Cell Tumor
Acronym: PAMSARC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Richard F Schlenk, Prof. Dr. med. Richard F. Schlenk (Coordinating Investigator), University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAMSARC
Record Dates: First submitted 2024-05-22; First posted 2024-06-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Desmoplastic Small Round Cell Tumor; Synovial Sarcoma
Keywords: SSTR; somatostatin receptor; SSTR2, SSTR3, SSTR5; somatostatin analog; pasireotide; fusion-gene driven; SS18-SSX1, SS18-SSX2, SS18-SSX4; EWSR1-WT1; extremely rare, aggressive sarcoma; maintaince therapy
MeSH Terms: conditions — Desmoplastic Small Round Cell Tumor; Sarcoma, Synovial | interventions — pasireotide

STUDY DESIGN:
Intervention Model Description: This is a single arm prospective, open label, multi-centre phase II study of pasireoide maintenance therapy in patients with advanced/metastatic DSRCT and SySa. According to the staggered approach during a run-in phase feasibility is assessed in 3 (or, if necessary, more) adult patients before initiating recruitment in adolescents. Adults receive 60 mg via intragluteal depot injection every 28±3 days, adolescents 60 mg (body surface area [BSA] >1.6 m²) or 40 mg (BSA 1.1-1.6 m2) via intragluteal depot injection every 28±3 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pasireotid treatment single arm (Experimental): Adults receive 60 mg via intragluteal depot injection every 28±3 days, adolescents 60 mg (body surface area [BSA] >1.6 m²) or 40 mg (BSA 1.1-1.6 m2) via intragluteal depot injection every 28±3 days.
  Interventions: Drug: Signifor

INTERVENTIONS:
Drug: Signifor — Signifor 40 mg: each vial contains 40 mg pasireotide (as pasireotide pamoate). Signifor 60 mg: each vial contains 60 mg pasireotide (as pasireotide pamoate).
  Other Names: ATC-Code: H01CB05

SUMMARY:
PAMSARC is a non-commercial interventional Phase 2 clinical trial of academic research institutions, with its primary goal being to improve medical treatment of fusion driven Desmoplastic small round cell tumor (DSRCT) and Synovial sarcoma (SySa) in young adults and adolsecents with male predominance.

Current management of DSRCT and SySa includes chemotherapy, radiation and aggressive cytoreductive surgery. Despite advances in multimodal therapy, outcomes remain poor with frequent disease recurrence and very limited options for patients with advanced disease.

Selected somatostatin receptor (SSTR) family members, i.e., SSTR2, SSTR3 and SSTR5, are frequently overexpressed in DSRCT and SySa, providing the rationale for treatment with somatostatin analogues (SSA).

Pasireotide is a SSA with high affinity for SSTR1, -2, -3, and -5 and is approved for the treatment of Cushing's disease and acromegaly and has also shown activity in other cancers. In patients with advanced stage DSRCT and SySa, conventional chemotherapeutic approaches frequently lead to disease response, however, the duration of progression-free time after chemotherapy is short. The targeted approach with pasireotide after initial intensive multimodal treatment may have the potential to significantly improve outcome.

DETAILED DESCRIPTION:
Desmoplastic small round cell tumor (DSRCT) is an extremely rare, aggressive sarcoma. It originates from the serosal surface of the abdominal cavity and the hallmark characteristic of DSRCT is the EWSR1-WT1 gene fusion. Synovial sarcoma (SySa) is also a rare fusion-gene driven (SS18-SSX1, SS18-SSX2, or rarely, SS18-SSX4) soft-tissue sarcoma.

Selected somatostatin receptor (SSTR) family members, i.e., SSTR2, SSTR3 and SSTR5, were highly expressed in patients with available transcriptome data, providing the basis for treatment with a somatostatin analog such as pasireotide with high affinity for SSTR1, 2, 3, and 5.

The primary aim of the study is to assess the clinical efficacy of pasireotide maintenance therapy for prolonging progression-free (PFS) and overall survival (OS) in patients with SSTR2/3/5-expressing advanced SySa and DSRCT. Furthermore measurable residual disease (MRD) before, during, and after pasireotide maintenance therapy are assessed. Pasireotide is applied in adults with 60 mg and in adolescents 60 mg (body surface area [BSA] >1.6 m²) or 40 mg (BSA 1.1-1.6 m²) via intragluteal via intragluteal depot injection every 28±3 days. The sample size is planned for the entire study population with subsequent sensitivity analysis in two subgroups, i.e., adolescents and adults. The primary efficacy analysis is be based on a two-sided, one-sample log-rank test using a significance level of 5%. The sample size was calculated assuming exponential data, planning for a power of 90% to detect a hazard ratio of 0.5. With a sample size of n=28, the expected number of events during the study is 22. Safety is assessed continuously according to CTCAE v5.0. The recruitment period is planned for 2 years starting in 2024 followed by a minimal follow-up of the last patient of 6 months leading to estimated trial completion in 2027.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting all of the following criteria are considered for enrolment into the trial:

1. Reference pathological proven diagnosis of DSRCT in any stage; or Reference pathological proven diagnosis of SySa, IRS III, metastatic or relapsed disease
2. High SSTR2/3/5 mRNA expression, as determined by RNA sequencing in the DKFZ/NCT/DKTK MASTER (ClinicalTrials.gov ID: NCT05852522) or INFORM programs.
3. Stable disease, partial or complete response after completion of standard treatment
4. Age from 13 to 50 years
5. For patients (≥16 years): Karnofsky-Index ≥ 80% For patients (<16 years): Lansky-Index ≥ 80%
6. No curative treatment option
7. Bodyweight ≥ 30kg and BSA ≥ 1.1m²
8. Time from last chemotherapy (at least 2 chemotherapy cycles) to enrollment <8 weeks
9. Ability of patient to understand character and individual consequences of the clinical trial
10. Written informed consent (for individuals <18 years of age an ICF for adolescents and their parents is needed)
11. For women of childbearing potential negative urine pregnancy test at screening as well as highly effective forms of contraception have to be in place thereafter

    * Evidence of childbearing potential is defined as fertile, following menarche and until becoming post-menopausal unless permanently sterile
    * Postmenopausal or evidence of non-childbearing status is defined as:

      * Amenorrhea for 1 year or more without an alternative medical cause following cessation of exogenous hormonal treatments plus follicle stimulating hormone (FSH) levels in the postmenopausal range in women not using hormonal contraception or hormonal replacement therapy.
      * Chemotherapy-induced menopause
      * Surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, total hysterectomy or tubal ligation at least 6 weeks before IMP treatment)
    * A man is considered fertile after puberty unless permanently sterile by bilateral orchidectomy
12. Female patients of childbearing potential and male patients with partners of childbearing potential who are sexually active must agree to the use of two forms of contraception in combination (male condom and one highly effective method). These should be started immediately after signing the informed consent form and continued throughout the period of study treatment plus 3 months for female and male patients . Male patients should refrain from fathering a child or donating sperm during the trial and for at least 3 months following the last dose.
13. Adequate bone marrow, renal, and hepatic function defined by laboratory tests within 14 days prior to study treatment:

    * Hemoglobin ≥ 10 g/dl
    * Neutrophil count ≥ 1,500/mm3
    * Platelet count ≥ 100,000/µl
    * Bilirubin ≤ 1.5 x upper limit of normal (ULN)
    * ALT and AST ≤ 2.5 x ULN
    * Alkaline phosphatase ≤ 2.5 x ULN
    * PT-INR/PTT ≤ 1.5 x ULN
    * Albumin ≥ 25 g/l
    * Creatine kinase ≤ 2.5 x ULN
    * Serum creatinine < or = 1.5 mg/dl or creatinine clearance = or > 51 ml/min (calculation according to Crockroft-Gault)

Exclusion Criteria:

Patients presenting with any of the following criteria are not included in the trial:

1. History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product
2. Concurrent or previous treatment within 30 days in another interventional clinical trial / Participation in other ongoing clinical trials.
3. Uncontrolled concurrent disease, in particular diabetes mellitus
4. Bleeding disorder
5. Therapeutic anticoagulation which cannot be paused temporarily in order to ensure safe intramuscular injection
6. Is taking or requiring any of the prohibited medication listed in Table 5 (6.4.2)
7. Heart rate at rest < 60/min
8. fasting glucose level > 110mg/dl
9. Severe neurologic or psychiatric disorder
10. Pregnancy/lactation
11. Prior treatment with somatostatin analog

    -

Ages: 13 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | PFS, measured from study registration to radiologically confirmed disease progression according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1, or death from any cause, whichever occurs first up to 4 years
  Assessment of clinical efficacy of pasireotide maintenance therapy

SECONDARY OUTCOMES:
overall survival (OS) | OS, measured from study registration to death from any cause (censoring of patients without an event at date of last follow-up) up to 4 years
  Assessment of clinical efficacy of pasireotide maintenance therapy

OTHER OUTCOMES:
measurable residual disease (MRD) | MRD before, during, and after pasireotide maintenance therapy up to 4 years
  Assessment of MRD and identify resistance mechanisms in liquid biopsies before, during, and after pasireotide maintenance therapy

CONTACTS AND LOCATIONS:
Overall Officials: Richard F. Schlenk, Professor, Principal Investigator — National Center for Tumour Diseases, University Hospital Heidelberg
Locations (4):
- Germany (4):
  - National Center for Tumour Diseases, University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg
  - Klinikum Stuttgart- Olga Hospital Zentrum für Kinder-, Jugend und Frauenmedizin, Stuttgart, Baden-Wurttemberg
  - Klinikum Stuttgart Studienzentrale Stuttgart Cancer Center, Tumorzentrum Eva-Mayr-Stihl, Stuttgart, Baden-Wurttemberg
  - Universitätsklinikum Essen Pädiatrische Hämatologie und Onkologie, Essen, North Rhine-Westphalia

REFERENCES:
- [Derived] Heilig CE, Heining C, Gnutzmann E, Roldan S, Heiligenthal L, Sparber-Sauer M, Hahn D, Dirksen U, Hamacher R, Florcken A, Thorwarth A, Deinzer CKW, Gaidzik VI, Pfaff E, Hubschmann D, Arndt K, Pfister SM, Glimm H, Frohling S, Schlenk RF. Rationale and design of the PAMSARC (pasireotide as maintenance treatment with monthly deep intramuscular injection in SSTR2/3/5-expressing synovial sarcoma and desmoplastic small round cell tumor) multicenter phase 2 trial. Cancer Treat Res Commun. 2025;45:100986. doi: 10.1016/j.ctarc.2025.100986. Epub 2025 Sep 3. PMID 40934647